CLINICAL TRIAL: NCT06965998
Title: A Pilot Randomized Double-Blinded Comparison of Full Treatment Dose Rivaroxaban for 90 Days to Prophylactic Dose Rivaroxaban for 45 Days in Patients With Lower Extremity Superficial Vein Thrombosis
Brief Title: A Pilot Trial Comparing Full Dose Rivaroxaban to Prophylactic Dose Rivaroxaban in Patients With Superficial Vein Thrombosis in the Leg
Acronym: RIVA-SVT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIVA-SVT Pilot
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: SVT; Thrombosis; Superficial Vein Thrombosis
Keywords: Pilot; Rivaroxaban; Feasibility; Full dose rivaroxaban; Treatment dose rivaroxaban; Superficial vein thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Intervention) (Experimental): Day 1-21: 15mg Rivaroxaban twice per day Day 22-90: 20mg Rivaroxaban once a day for 69 days
  Interventions: Drug: Full dose rivaroxaban
- Group B (Comparator) (Active Comparator): Day 1-21: 10mg Rivaroxaban once a day AND placebo once a day Day 22-45: 10mg Rivaroxaban once a day Day 46-90: Placebo once a day for 45 days
  Interventions: Drug: Low dose rivaroxaban; Drug: Placebo

INTERVENTIONS:
Drug: Full dose rivaroxaban — The intervention group will receive full dose rivaroxaban for 90 days.
  Arms: Group A (Intervention)
Drug: Low dose rivaroxaban — The comparator group will receive the standard treatment of low dose rivaroxaban.
  Arms: Group B (Comparator)
Drug: Placebo — Since the treatment arm has an AM and PM dose of study drug from Day 1-21, the comparator group will take 1 placebo pill in the PM to keep the two arms blinded.
  Arms: Group B (Comparator)

SUMMARY:
The goal of this clinical trial, called a pilot study or a feasibility study, is to test the study plan and to find out whether enough participants will join a larger study and accept the study procedures. This type of study includes a small number of participants so it is not expected to prove how safe the treatment is or how well the treatment works.

The main question it hopes to answer is:

1.What is the average number of patients that are recruited per month during the 12 month study period?

To test the study plan, adults being treated for a superficial vein thrombosis (SVT), which is a blood clot in the superficial veins of the leg, will be given a type of blood thinner called rivaroxaban. Half of the participants in this study will be given the standard (low-dose) rivaroxaban for 45 days, then 45 days of placebo (a substance that looks like the study medication but does not have any active or medicinal ingredients). The other half of participants will be given full-dose rivaroxaban for a total of 90 days. The placebo in this study is not intended to have any effect on the participants blood clot. A placebo is used to make the results of the study more reliable.

DETAILED DESCRIPTION:
The standard or usual treatment for a superficial vein thrombosis (SVT) is to treat with a low-dose (often called a prophylactic dose) of blood thinner for 45 days. Rivaroxaban is a type of oral blood thinner that is used in the treatment and prevention of blood clots. Currently, rivaroxaban 10mg daily for 45 days is the most commonly used treatment in patients with lower extremity SVT.

Recent studies of participants with SVT suggest that treatment with full-dose (sometimes called therapeutic dose) blood thinners could be promising in preventing additional complications from SVT such as:

* A new blood clot in the deep veins of the legs or arms
* A new pulmonary embolism (a blood clot in the lungs)
* A recurrence or extension of the existing SVT (the existing clot comes back after treatment is stopped or gets bigger)

The Investigators are studying whether a full-dose of rivaroxaban for 90 days could prevent or improve additional complications from SVT.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age ≥ 18 years old.
2. Objectively confirmed diagnosis within 14 days of an acute symptomatic SVT of the lower extremities by standardized CUS, where SVT is defined as incompressibility of a venous segment located along the course of a known superficial vein.
3. Anticoagulation for SVT is warranted per clinicians.
4. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Other indication(s) for therapeutic or prophylactic dose anticoagulation (e.g. atrial fibrillation, mechanical valve, etc.).
2. History of PE or DVT within 6 months (180 days) of screening.
3. >5 days of any anticoagulants for the index SVT.
4. Requires use of aspirin >100mg daily or other antiplatelet agents.
5. Patients receiving concomitant systemic treatment with strong inhibitors of both CYP 3A4 and P-gp (e.g. cobicistat, ketoconazole, itraconazole, posaconazole, ritanovir, etc.).
6. Active bleeding or history of CRNMB or major bleeding (as defined by the ISTH) within 30 days of screening.
7. History of severe head trauma or ophthalmic, spinal, cerebral surgery within 90 days of screening.
8. Have acute endocarditis.
9. Thrombocytopenia (platelet count <50,000/uL), acute hepatitis, chronic active hepatitis, cirrhosis with severe hepatic impairment defined by a Childs-Pugh class B or C.
10. Creatinine clearance <30 ml/min.
11. Known contraindication to treatment with rivaroxaban.
12. Are participating in another interventional trial that would compromise the results or integrity of this trial as determined by the investigator.
13. Pregnant or breast feeding.
14. Known hereditary or acquired severe hemorrhagic disease.
15. Life expectancy <3 months.
16. Unstable medical or psychological condition that would interfere with trial participation at the discretion of the site investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Outcome | 12 months from when recruitment opens.
  The primary feasibility outcome of this pilot trial is the average number of patients recruited per month during the 12 month recruitment period.

SECONDARY OUTCOMES:
Secondary Feasibility Outcomes | From the start of study recruitment to the last follow-up of the last participant enrolled.
  The rate (%) of eligible patients that give consent to participate.
Secondary Feasibility Outcomes | From the start of study recruitment to the last follow-up of the last participant enrolled.
  The rate (%) of patients that are not lost to follow-up.
Secondary Feasibility Outcomes | From the start of study recruitment to the last follow-up of the last participant enrolled.
  The rate (%) of patients who complete and adhere to the study procedures.
Secondary Feasibility Outcomes | From the start of study recruitment to the last follow-up of the last participant enrolled.
  Reasons why eligible patients chose not to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Fei Wang, MD,MPH, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital Montfort, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyer-Westendorf J, Schellong SM, Gerlach H, Rabe E, Weitz JI, Jersemann K, Sahin K, Bauersachs R; SURPRISE investigators. Prevention of thromboembolic complications in patients with superficial-vein thrombosis given rivaroxaban or fondaparinux: the open-label, randomised, non-inferiority SURPRISE phase 3b trial. Lancet Haematol. 2017 Mar;4(3):e105-e113. doi: 10.1016/S2352-3026(17)30014-5. Epub 2017 Feb 16. PMID 28219692
- [Background] Samama MM. The mechanism of action of rivaroxaban--an oral, direct Factor Xa inhibitor--compared with other anticoagulants. Thromb Res. 2011 Jun;127(6):497-504. doi: 10.1016/j.thromres.2010.09.008. Epub 2010 Oct 2. PMID 20888031
- [Background] Blondon M, Righini M, Bounameaux H, Veenstra DL. Fondaparinux for isolated superficial vein thrombosis of the legs: a cost-effectiveness analysis. Chest. 2012 Feb;141(2):321-329. doi: 10.1378/chest.11-0625. Epub 2011 Jul 14. PMID 21757569
- [Background] Wichers IM, Di Nisio M, Buller HR, Middeldorp S. Treatment of superficial vein thrombosis to prevent deep vein thrombosis and pulmonary embolism: a systematic review. Haematologica. 2005 May;90(5):672-7. PMID 15921382
- [Background] Duffett L. Management of Superficial Venous Thrombosis: A Systematic Review of Literature and Survey of Canadian Physicians. Thesis. Université d'Ottawa / University of Ottawa; 2018. doi:10.20381/ruor-21377
- [Background] Duffett L, Kearon C, Rodger M, Carrier M. Treatment of Superficial Vein Thrombosis: A Systematic Review and Meta-Analysis. Thromb Haemost. 2019 Mar;119(3):479-489. doi: 10.1055/s-0039-1677793. Epub 2019 Feb 4. PMID 30716777
- [Background] Frappe P, Buchmuller-Cordier A, Bertoletti L, Bonithon-Kopp C, Couzan S, Lafond P, Leizorovicz A, Merah A, Presles E, Preynat P, Tardy B, Decousus H; STEPH Study Group. Annual diagnosis rate of superficial vein thrombosis of the lower limbs: the STEPH community-based study. J Thromb Haemost. 2014 Jun;12(6):831-8. doi: 10.1111/jth.12575. PMID 24679145
- [Background] Leon L, Giannoukas AD, Dodd D, Chan P, Labropoulos N. Clinical significance of superficial vein thrombosis. Eur J Vasc Endovasc Surg. 2005 Jan;29(1):10-7. doi: 10.1016/j.ejvs.2004.09.021. PMID 15570265
- [Background] Di Minno MN, Ambrosino P, Ambrosini F, Tremoli E, Di Minno G, Dentali F. Prevalence of deep vein thrombosis and pulmonary embolism in patients with superficial vein thrombosis: a systematic review and meta-analysis. J Thromb Haemost. 2016 May;14(5):964-72. doi: 10.1111/jth.13279. Epub 2016 Mar 15. PMID 26845754
- [Background] Di Nisio M, Wichers IM, Middeldorp S. Treatment for superficial thrombophlebitis of the leg. Cochrane Database Syst Rev. 2018 Feb 25;2(2):CD004982. doi: 10.1002/14651858.CD004982.pub6. PMID 29478266
- [Background] Geersing GJ, Cazemier S, Rutten F, Fitzmaurice DA, Hoes AW. Incidence of superficial venous thrombosis in primary care and risk of subsequent venous thromboembolic sequelae: a retrospective cohort study performed with routine healthcare data from the Netherlands. BMJ Open. 2018 Apr 20;8(4):e019967. doi: 10.1136/bmjopen-2017-019967. PMID 29678975
- [Background] Beyer-Westendorf J. Controversies in venous thromboembolism: to treat or not to treat superficial vein thrombosis. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):223-230. doi: 10.1182/asheducation-2017.1.223. PMID 29222259
- [Background] Bauer KA, Hawkins DW, Peters PC, Petitou M, Herbert JM, van Boeckel CA, Meuleman DG. Fondaparinux, a synthetic pentasaccharide: the first in a new class of antithrombotic agents - the selective factor Xa inhibitors. Cardiovasc Drug Rev. 2002 Winter;20(1):37-52. doi: 10.1111/j.1527-3466.2002.tb00081.x. PMID 12070533
- [Background] Mathieu ME, Duffett L, Caiano L, Scarvelis D, Code C, Wells P, Le Gal G. Management and outcomes of superficial vein thrombosis: a single-center retrospective study. Res Pract Thromb Haemost. 2023 Nov 18;8(1):102263. doi: 10.1016/j.rpth.2023.102263. eCollection 2024 Jan. PMID 38187826